CLINICAL TRIAL: NCT04715022
Title: Sympathetic-vascular Dysfunction in Obesity and Insulin Resistance
Brief Title: Sympathetic-vascular Dysfunction in Obesity and Insulin Resistance (Vitamin C Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Holwerda PhD, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00146744
Record Dates: First submitted 2021-01-10; First posted 2021-01-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo infusion (Placebo Comparator): Saline will be administered over 2 hours
  Interventions: Drug: Saline
- Ascorbic acid infusion (Active Comparator): Ascorbic acid solution (American Regent Laboratories Inc.) will be obtained from the KU Investigational Pharmacy located in the University of Kansas (KU) Clinical Research Center where studies will take place. A priming bolus of 0.06 g ascorbic acid/kg fat free mass (FFM) dissolved in 100 mL of saline will be infused intravenously at 5 mL/min for 20 minutes, followed immediately by a "drip-infusion" of 0.02 g/kg FFM dissolved in 30 mL of saline administered over 2 hours at 0.5 mL/min.
  Interventions: Drug: Ascorbic acid solution (American Regent Laboratories Inc.)

INTERVENTIONS:
Drug: Ascorbic acid solution (American Regent Laboratories Inc.) — Ascorbic acid solution (American Regent Laboratories Inc.) will be obtained from the KU Investigational Pharmacy located in the KU Clinical Research Center where studies will take place. A priming bolus of 0.06 g ascorbic acid/kg fat free mass (FFM) dissolved in 100 mL of saline will be infused intravenously at 5 mL/min for 20 minutes, followed immediately by a "drip-infusion" of 0.02 g/kg FFM dissolved in 30 mL of saline administered over 2 hours at 0.5 mL/min.
  Arms: Ascorbic acid infusion
Drug: Saline — Placebo (saline) will be administered
  Arms: Placebo infusion

SUMMARY:
The main purpose of research is to examine and understanding the development of hypertension in obese adults with insulin resistance. Findings from our studies will identify unique mechanisms that can be targeted to limit increases in vascular dysfunction and reduce the excessively high prevalence of hypertension and risk for cardiovascular disease (CVD).

This study is testing the health of the blood vessels and the activity of the nerves that control the blood vessels in adults with insulin resistance. The extent to which ascorbic acid (Vitamin C) improves the function of the blood vessels will be determined. The primary outcome is blood pressure, which is the result of blood vessel health and activity of the nerves, and the reduction in blood pressure that is observed with ascorbic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Obese: BMI >30 m/kg2
2. Middle-aged: 35-65 years
3. Participants must be willing and able to discontinue taking any vitamin C or E supplements or omega-3 fatty acids beginning 2 weeks prior.
4. Able and willing to provide written informed consent

Exclusion Criteria:

1. Diabetes mellitus: fasting glucose < 1267 mg/dL and/or HbA1c < 6.5%
2. Currently taking a statin or antihypertension medication
3. Hyperlipidemia: Fasting triglycerides < 250 mg/dL
4. Hypertension: <130/80 mmHg
5. History of heart disease (e.g., myocardial infarction, stent)
6. History of vascular disease (e.g., bypass, stroke)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of infusion of ascorbic acid | 30 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of infusion of ascorbic acid | 60 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of infusion of ascorbic acid | 90 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of infusion of ascorbic acid | 120 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Holwerda, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No